CLINICAL TRIAL: NCT01231763
Title: Film Acceptability Characterization and Evaluation
Brief Title: Acceptability Study of Vaginal Films for HIV Prevention
Acronym: FACE
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sharon Hillier, PhD, University of Pittsburgh
Other Study IDs: PRO10080621 (UPittsburgh IRB#)
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections; Anti-Infective Agents
Keywords: HIV prevention; Vaginal film; Microbicide; Administration, intravaginal
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers
  Interventions: Other: No intervention (not applicable)

INTERVENTIONS:
Other: No intervention (not applicable) — No intervention (not applicable)

SUMMARY:
This study is being done to find out what women would want in a film vaginal product for human immunodeficiency virus (HIV) prevention, especially what it should look like and how to apply it.

The investigators hypothesize that women will prefer a smooth, clear, and rectangular quick-dissolve vaginal film for HIV prevention over a textured, opaque, square quick-dissolve vaginal film.

DETAILED DESCRIPTION:
The lives of 25 million people have ended due to HIV-related causes since the start of the AIDS epidemic in 1981 (1). Each year, AIDS continues to claim the lives of millions of people, with an estimated two million deaths worldwide in 2008 (2). Heterosexual transmission of HIV accounts for the majority of new infections and disproportionately affects women both in the United States and globally (2, 3). There is an urgent need for agents to prevent the sexual transmission of HIV, particularly agents that may be controlled by women.

Quick dissolve films such as Listerene® Breath Strips have been developed for inexpensive delivery of drugs and vitamins. As products for HIV prevention, quick dissolve films offer a host of potential advantages including low cost, control by the receptive partner, discreet and applicator-free use, low mess, portability, easy storage, stability, targeting to site of exposure, reduction of systemic toxicity by bypassing first-pass metabolism, and the incorporation of multiple active microbicidal compounds (4, 5).

In the course of developing agents for HIV prevention, determination of valued characteristics is important for product refinement and for enhancement of future use likelihood. Knowledge regarding acceptability can also inform product promotion and educational campaigns (6).

ELIGIBILITY:
Inclusion Criteria:

* Female 18-30 years old at time of enrollment
* Able to provide written informed consent

Exclusion Criteria:

* Not sexually active, defined as no vaginal sex at any time in the past year
* Pregnant by self-report

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18-30 years from the Pittsburgh, Pennsylvania area who express interest in the study. Enrollment is expected to achieve racial and ethnic demographics representative of Allegheny County, Pennsylvania in terms of approximately 0.2 percent American Indian and Alaska Native, 2.5 percent Asian, and 1.5 percent Hispanic or Latino (7). Allegheny County is 82.8 percent white and 13.2 percent black or African American (7). For enrollment in this study, we would like to achieve at least 40 percent black or African American in order to collect a more diverse set of film microbicide preferences. The remainder of enrollment is expected to be white.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Preferred physical characteristics of a vaginal film product | One visit lasting two hours
  Preferred texture, shape, size, and appearance of a vaginal film product via focus group discussion and questionnaires

SECONDARY OUTCOMES:
Valued vaginal product characteristics | One visit lasting two hours
  Desired characteristics of vaginal products such as lubrication, prescription status, and contraceptive function via focus group discussion and questionnaires
Impressions regarding vaginal films | One visit lasting two hours
  Impressions about vaginal films such as ease of use, comfort, and effect on sexual pleasure via focus group discussion and questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Magee-Womens Research Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Joint United Nations Programme on HIV/AIDS. 08 Report on the global AIDS epidemic. 2008 Available from: http://www.unaids.org/en/KnowledgeCentre/HIVData/GlobalReport/2008/2008_Global_report.asp.
- [Background] Joint United Nations Programme on AIDS, WHO. AIDS Epidemic Update. 2009 Available from: http://data.unaids.org/pub/Report/2009/JC1700_Epi_Update_2009_en.pdf.
- [Background] Centers for Disease Control and Prevention (CDC). Subpopulation estimates from the HIV incidence surveillance system--United States, 2006. MMWR Morb Mortal Wkly Rep. 2008 Sep 12;57(36):985-9. PMID 18784639
- [Background] Sassi AB, McCullough KD, Cost MR, Hillier SL, Rohan LC. Permeability of tritiated water through human cervical and vaginal tissue. J Pharm Sci. 2004 Aug;93(8):2009-16. doi: 10.1002/jps.20107. PMID 15236450
- [Background] Romano J, Malcolm RK, Garg S, Rohan LC, Kaptur PE. Microbicide delivery: formulation technologies and strategies. Curr Opin HIV AIDS. 2008 Sep;3(5):558-66. doi: 10.1097/COH.0b013e328305b96e. PMID 19373022
- [Background] Mantell JE, Myer L, Carballo-Dieguez A, Stein Z, Ramjee G, Morar NS, Harrison PF. Microbicide acceptability research: current approaches and future directions. Soc Sci Med. 2005 Jan;60(2):319-30. doi: 10.1016/j.socscimed.2004.05.011. PMID 15522488
- [Background] U.S. Census Bureau. Allegheny County QuickFacts. [updated 4-22-2010]; Available from: http://quickfacts.census.gov/qfd/states/42/42003.html.